CLINICAL TRIAL: NCT02056210
Title: Mobilization Test of BM Progenitor Cells With Plerixafor / AMD3100: Controlled Parallel Group Comparison Between Diabetic and Non Diabetic Subjects
Brief Title: Stem Cell Mobilization With Plerixafor in Diabetic vs Control Subjects
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Padova (Other)
Collaborators: Azienda Ospedaliera di Padova (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MZBL-2996P/13
Record Dates: First submitted 2014-02-03; First posted 2014-02-05 (Estimated); Last update posted 2014-10-24 (Estimated); Status verified 2014-10

CONDITIONS: Diabetes
Keywords: Stem cells; Bone marrow
MeSH Terms: conditions — Diabetes Mellitus | interventions — plerixafor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Stem cell mobilization in diabetic patients (Experimental): Injection of Mozobil (Plerixafor / AMD3100) in diabetic patients
  Interventions: Drug: Mozobil
- Stem cell mobilization in non diabetic subjects (Experimental): Injection of Mozobil (Plerixafor / AMD3100) in non diabetic subjects
  Interventions: Drug: Mozobil

INTERVENTIONS:
Drug: Mozobil — Subcutaneous injection of 0.24 mg/kg Mozobil once at 8:30am
  Other Names: Plerixafor; AMD3100

SUMMARY:
The objective of this study is to assess whether there are differences in the mobilization of CD34+ cells and EPC in response to Mozobil in patients with diabetes mellitus compared to subjects without diabetes. Currently, there are no non-invasive methods for the study of bone marrow function in humans. This project aims to evaluate in patients with type 1 or type 2 diabetes mellitus the ability to mobilize CD34+ cells and EPC from the bone marrow to the periphery in response to the exogenous mobilizing agent AMD3100 / plerixafor (Mozobil), compared with a group of non-diabetic individuals. While it has been recently shown that diabetic patients do not respond to mobilization induced by G-CSF (Filgrastim), the investigators herein hypothesize that diabetic patients can adequately respond to mobilization induced by Plerixafor

DETAILED DESCRIPTION:
Scientific background. Diabetes mellitus is associated with an increased prevalence and incidence of cardiovascular diseases. It is believed that the high cardiovascular risk in diabetes is attributable to the adverse effects of glucotoxicity and lipotoxicity on endothelial cells. Recent data indicate that endothelial repair mechanisms play an important role in determining the integrity of the endothelium and thus the global health of the cardiovascular system. Data from our research group demonstrated that the cells involved in endothelial regeneration and neo-angiogenesis (including CD34+ cells and endothelial progenitor cells, EPC) are reduced in number and dysfunctional in patients with diabetes mellitus. EPC belong to the CD34+ cell population and are defined based on the co-expression of endothelial-lineage markers, such as VEGF receptor 2 (VEGFR2 or KDR). These cells are further impaired in diabetic patients with cardiovascular disease. It is believed that these changes represent one of the causes of cardiovascular damage in diabetes.

The mechanisms underlying the decrease of EPC and other progenitor cells in diabetes are not fully understood. Normally, EPC reside in the bone marrow and their circulating levels in peripheral blood are very low. In response to ischemic injury or vascular damage, EPC are mobilized from the bone marrow to peripheral blood. Data obtained in experimental models of diabetes mellitus indicate a defect in EPC mobilization from the bone marrow to the peripheral circulation in response to ischemia, which results in an impairment of the post-ischemic neo-angiogenetic processes. Similar experimental results were obtained by different research groups. Our data also show that experimental diabetes reduces the marrow response to exogenous mobilizing agents such as G-CSF and SCF. Other clinical data in humans from our and other research groups confirm the hypothesis of a defect in the bone marrow of patients with diabetes mellitus. In particular, diabetes causes profound alterations of the bone marrow microenvironment associated with microangiopathy and alteration of the stem cells niche. These results confirm a study in the mouse model of type 1 diabetes, in which it was for the first time identified a specific form of microangiopathy causing depletion of CD34+ cells and EPC in the bone marrow.

As a consequence of this bone marrow damage, our research group has recently shown that the mobilization of CD34+ cells and EPC phenotypes is profoundly defective in patients with type 1 and 2 diabetes mellitus.

To reach this conclusion, the investigators used a test of bone marrow reserve by administering low dose human recombinant G-CSF (Filgrastim). The study showed that a sub-maximal marrow stimulation is able to highlight differences between diabetics and non-diabetics and is absolutely safe, since there have been no significant side effects. In a hematology context, it was also previously shown that diabetes is a factor predictive of "poor mobilization" exposing patients to an increased risk of failing stem cell collection for autologous stem cell transplantation.

From a functional/mechanistic standpoint, it has been demonstrated that an impairment of the CXCL12/CXCR4 axis probably contributes to the lack of mobilization of bone marrow stem/progenitor cells associated with diabetes. The drug AMD3100 / plerixafor (Mozobil ®) is a direct antagonist of CXCR4 and inhibits the cellular signal keeping stem / progenitor cells within the bone marrow. For this reason, AMD3100 / Plerixafor is rapidly effective for the mobilization of bone marrow stem cells. From an experimental point of view, it was observed that diabetic animals, although not responsive to mobilization induced by ischemia and G-CSF, are responsive to mobilization induced by AMD3100 / Plerixafor. Mozobil is currently approved in Italy for stem cell mobilization in patients with multiple myeloma or lymphoma for the purpose of auto-transplantation, in combination with G-CSF, in poorly mobilizing patients (see SmPC). At this stage, the effectiveness of Mozobil in inducing mobilization of stem / progenitor cells in diabetic patients has not yet been tested.

Scientific question. The objective of this study is to assess whether there are differences in the mobilization of CD34+ cells and EPC in response to Mozobil in patients with diabetes mellitus compared to subjects without diabetes. Currently, there are no non-invasive methods for the study of bone marrow function in humans. This project aims to evaluate in patients with type 1 or type 2 diabetes mellitus the ability to mobilize CD34+ cells and EPC from the bone marrow to the periphery in response to the exogenous mobilizing agent AMD3100 / plerixafor (Mozobil), compared with a group of non-diabetic individuals. While it has been recently shown that diabetic patients do not respond to mobilization induced by G-CSF (Filgrastim), the investigators herein hypothesize that diabetic patients can adequately respond to mobilization induced by Plerixafor.

Plausibility and clinical relevance. It is believed that alterations of stem/progenitor cells secondary to a bone marrow defect contribute to the development of clinical diabetic microangiopathy and macroangiopathy. For this reason, it is of great interest to explore the mechanisms causing an progenitor cell defects in diabetes and the possible strategies to cope with this. A wealth of data coming from animal, human and epidemiologic studies indicate that the mobilizing response to G-CSF is impaired in diabetic patients. Therefore, stem mobilization in diabetes has to be considered an "unmet clinical need". On the other side, preclinical experimental data in animal models of diabetes indicate that AMD3100 / Plerixafor is able to mobilize stem and progenitor cells. The clinical relevance of the project lies in the possibility to identify a treatment able to restore stem/progenitor cell mobilization in diabetes. This can have favorable implications for chronic diabetic complications, such as microangiopathy and cardiovascular diseases. In fact, this project is relevant from a pathophysiological point of view, since it is believed that EPC should protect against vascular complications of diabetes. Furthermore, from a hematologic standpoint, being aware that diabetic patients are hyporesponsive to G-CSF whilst responding adequately to Plerixafor would allow to individualize mobilization protocols in view of an autologous hematopoietic stem cell transplantation.

Expected adverse events. Treatment with Mozobil in combination with G-CSF may be associated with mild adverse events (see SmPC). Compared to placebo + G-CSF, the use of Mozobil + G-CSF in patients from two clinical trials induced a significantly higher number of grade 1-2 adverse reactions: diarrhea (37% vs 17%), nausea (34% vs 22%), flatulence (7% vs 3%), injection site reactions (34% vs 10%), dizziness (11% vs 6%). No side effects of grade 3-4 were reported.

In the present study Mozobil will be given as monotherapy, ie not in combination with G-CSF. Based on literature data, adverse events that may be expected with this type of treatment are mild:

* In a study of 20 healthy volunteers grade 1 side effects were reported in response to a monotherapy treatment with Mozobil sc: cramps or bloating, flatulence, dry mouth.
* In a study that involved 10 healthy volunteers treated with Mozobil sc monotherapy the following mild side effects were observed (grade 1): erythema or itching at the site of injection, headache, perioral paresthesia, nausea, abdominal swelling.
* A study that involved 25 healthy donors treated with Mozobil sc monotherapy reported the following adverse events of grade 1 (mild): dizziness, nausea, flatulence, discomfort or feeling of warmth at the injection site, perioral paresthesias, sweating, cephalea.

On the basis of these data, it can be assumed that the use of Mozobil monotherapy is safe and expected side effects are mild and tolerable for the patient.

In addition, as with almost all drugs, Mozobil can induce allergic reactions and anaphylaxis.

ELIGIBILITY:
Inclusion criteria:

* Diabetes mellitus (type 1 or 2) (for the patients) or absence of diabetes mellitus and other carbohydrates metabolism alterations (for the non diabetic controls)
* Age 20-65 years;
* Both genders;
* Informed consent.

Exclusion criteria:

* Age <20 or >65 years;
* Pregnancy or lactation *
* Recent surgery or trauma;
* Recent acute diseases (within 2 months from study entry);
* Immune diseases (except from type I diabetes and autoimmune thyroiditis);
* Chronic infectious diseases;
* Hematologic malignancies either past or present;
* Solid tumor known or strongly suspected;
* Leukocytosis, leukopenia, or thrombocytopenia;
* Solid organ transplant or immunosuppression;
* Alteration of hepatic function (transaminases >2 ULN);
* Severe chronic diabetic micro- or macroangiopathy
* HbA1c >11%.
* Deficit in renal function (eGFR<50 ml/m2);
* Significant abnormalities of the peripheral lymphocyte immunophenotype;
* Known hypersensitivity to Mozobil or its excipients;
* Refusal / inability to provide informed consent.

  * women with childbearing potential can participate to this trial just if are using effective oral contraception; a negative pregnancy test is required before study entry). Women will be asked to continue oral contraception for 3 months after Mozobil administration.

All antidiabetic medications are allowed.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2014-02; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
CD34+ stem cell mobilization in diabetic vs non diabetic subjects | 6 hours
  To evaluate the differences of CD34+ cells mobilization from the bone marrow to the peripheral blood induced by a single sc injection of Mozobil in diabetic patients versus non diabetic controls.
  Clinical response variable: comparison of the fold change in CD34+ peripheral cell count in diabetic versus non diabetic controls after Mozobil administration (with collection of safety and tolerability data).

SECONDARY OUTCOMES:
CD34+ stem cell mobilization within diabetic patients | 6 hours
  to evaluate whether Mozobil monotherapy is able to induce a significant CD34+ stem cells mobilization in diabetic patients (intra-group comparison).
  Clinical response variable: detection of a significant fold-change in CD34+ peripheral cell count versus baseline in diabetic patients.
EPC (endothelial progenitor cell) mobilization in diabetic vs non diabetic subjects | 6 hours
  To evaluate the differences in mobilization of EPC (CD34+KDR+) from the bone marrow to the peripheral blood induced by a single sc injection of Mozobil in diabetic patients versus non diabetic controls (inter-group comparison).
  Clinical response variable: comparison of the fold change in CD34+ KDR+ peripheral cell count in diabetic versus non diabetic controls after Mozobil administration (with collection of safety and tolerability data).
EPC (endothelial progenitor cell) mobilization within diabetic patients | 6 hours
  To evaluate whether Mozobil monotherapy is able to induce a significant EPC mobilization in diabetic patients (intra-group comparison).
  Clinical response variable: detection of a significant fold-change in CD34+KDR+ peripheral cell count versus baseline in diabetic patients

CONTACTS AND LOCATIONS:
Locations (1):
- Policlinico Universitario, Azienda Ospedaliera di Padova, Padua, Italy

REFERENCES:
- [Derived] Fadini GP, Fiala M, Cappellari R, Danna M, Park S, Poncina N, Menegazzo L, Albiero M, DiPersio J, Stockerl-Goldstein K, Avogaro A. Diabetes Limits Stem Cell Mobilization Following G-CSF but Not Plerixafor. Diabetes. 2015 Aug;64(8):2969-77. doi: 10.2337/db15-0077. Epub 2015 Mar 24. PMID 25804941